CLINICAL TRIAL: NCT03660215
Title: Interventional Trial in Primary Care of Medico-social Mediation on the Prevention of the Return to Emergencies Among People in a Precarious Social Situation
Brief Title: Medico-social Mediation on the Prevention of the Return to Emergencies Among People in a Precarious Social Situation
Acronym: M2PRUSSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-08
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Social Isolation
MeSH Terms: conditions — Social Isolation | interventions — Mediation Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): usual charge
- experimental group (Experimental): Mediation:
  The mediator will intervene on several levels: planning of care according to the medical prescriptions on a support adapted and comprehensible by the patient according to his level of health literacy and his linguistic capacities, coaching on the management of the chronic diseases, possible orientation towards a workshop of therapeutic education, appointments calendar, clear indication of treatment changes, provision of contact information for allied health professionals , assistance in making appointments, possible accompaniments at a professional health.
  Interventions: Other: mediation

INTERVENTIONS:
Other: mediation — support throughout their care journey during the 90 days following an emergency visit. This support will be carried out by a specific staff trained in medico-social mediation
  Arms: experimental group

SUMMARY:
This research aims to evaluate a new mode of care for precarious public through a medico-social mediation device after emergencies, with the aim of improving their care and to prevent possible complications.

The main objective is to evaluate the effectiveness of management by a medico-social mediation device set up within 48 hours after leaving emergency on the 90-day emergency readmission rate. people living in precarious situations.

prospective randomized interventional trial with two arms. Patients will complete questionnaires assessing precariousness, quality of life, health literacy, and time perspective. Eligible patients (726 subjects) are randomized : control group (usual management) or experimental group (patient is contacted within 48 hours by a medico-social mediator familiar with the territory), and followed for 90 days by the latter, in order to optimize and secure the care path.

Readmissions are identified from emergency database and Regional Emergency Terminal and documented.

Patients in the experimental group benefit from the support of a local health mediator who carries out a diagnosis of the person's needs in order to follow his or her care path in an optimal way. It implements and ensures with the patient and his entourage the follow-up of the care through his network of professionals of the social sector and the health.

The study will be under the responsibility of a multidisciplinary scientific committee experienced in public health, epidemiology and social psychology of health, in the field of emergencies, precariousness and medico-social mediation, and excellent knowledge. territories concerned.

DETAILED DESCRIPTION:
This research aims to evaluate a new mode of care for precarious public through a medico-social mediation device after emergencies, with the aim of improving their care, to prevent possible complications of diseases related to poor / no return home care, to improve the quality of life of the people concerned, and to participate in the decongestion of emergencies.

The main objective is to evaluate the effectiveness of management by a medico-social mediation device set up within 48 hours after leaving emergency on the 90-day emergency readmission rate. people living in precarious situations.

Secondary objectives:

* Evaluate the effectiveness of the studied CEP on the 180-day emergency readmission rate, the hospitalization rate at 30, 90 days and 180 days, the number of readmissions to emergencies within 30, 90 and 180 days of follow-up, duration of hospitalizations occurring within 180 days, subgroups of patients, reasons for readmissions to the emergency department,
* Evaluate the impact of health literacy and temporal awareness levels on the 90 day emergency readmission rate,
* Evaluate the impact of the initial quality of life on the 90-day readmission rate,
* Identify predictive factors for readmission to emergencies at 30, 90 and 180 days.

Methodological approach: prospective randomized interventional trial with two arms.

Patients admitted to one of the four participating UAs meeting the inclusion / exclusion criteria of the trial will complete questionnaires assessing precariousness, quality of life, health literacy, and time perspective. Two emergency centers will be located in dense urban areas that are highly vulnerable (Marseille's northern neighborhoods); two others in less urbanized areas in which there are pockets of neo-rural precariousness. Eligible patients are randomized to emergency in one of the two arms (control: usual management) or (experimental: intervention). In this last arm, the patient is contacted within 48 hours by a medico-social mediator familiar with the territory, and followed for 90 days by the latter, in order to optimize and secure the care path. Patients are recalled at 90 days (number obtained at the signing of the consent). Patients are documented for emergency use, severity (CCMU score), primary and associated conditions, quality of life (WHOQOL-Brief), patterns and patterns of discharge. A health literacy score and a time-domain assessment (short-term PTZ) will be administered only in the experimental arm, using these scales to cover a secondary objective to examine the impact of health literacy and literacy. temporal perspective on the readmission rate. Readmissions are identified from the emergency database and Regional Emergency Terminal and documented (reason for appeal, severity score, mode and reason for leaving the study).

Patients in the experimental group benefit from the support of a local health mediator who carries out a diagnosis of the person's needs in order to follow his or her care path in an optimal way. It implements and ensures with the patient and his entourage the follow-up of the care through his network of professionals of the social sector and the health.

Patients in the control group do not have the support of the health mediator. They are only initially evaluated. Their eventual readmission is identified from the local emergency database at 30, 90 and 180 days as patients in the experimental group.

The number of subjects needed to carry out the research is 726 subjects, ie 363 subjects per group.

The statistical analyzes are carried out according to an analysis plan validated by the scientific committee of the study, with robust tools , blind (with lifting of the blind at the end of the analyzes). Use of descriptive and then analytical techniques.

The study will be under the responsibility of a multidisciplinary scientific committee experienced in public health, epidemiology and social psychology of health, in the field of emergencies, precariousness and medico-social mediation, and excellent knowledge. territories concerned.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to emergencies,
* Social precariousness score at the EPICES scale,
* Having made at least one visit to an emergency department during the 90 days prior to inclusion,
* Arriving on their own or being transported to a recumbent position by firefighters or an ambulance,
* Volunteers to participate in the study ,

Exclusion Criteria:

Having a score of social precariousness according to the EPICES scale lower than 30, Transferred from a medico-social institution, Unable to answer a questionnaire, face-to-face with an interviewer, either for medical reasons Coming to emergencies for / with a psychiatric decompensation and / or presenting a serious mental illness and / or under the influence of psychotropes, Residing outside the areas of residence targeted by the research, Refusing to participate in the study , In situations of legal incapacity to fulfill informed consent, in particular persons under guardianship or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
numbers of readmission to hospital emergencies | 90 days
  90-day readmission rate to hospital emergencies

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France

REFERENCES:
- [Derived] Rotily M, Persico N, Lamouroux A, Rojas-Vergara AC, Loundou A, Boucekine M, Apostolidis T, Odena S, Chischportich C, Auquier P. Health mediation does not reduce the readmission rate of frequent users of emergency departments living in precarious conditions: what lessons can be learned from this randomised controlled trial? BMC Emerg Med. 2024 May 15;24(1):83. doi: 10.1186/s12873-024-01000-2. PMID 38750416